CLINICAL TRIAL: NCT04929912
Title: Electroporation for Cancer Treatment Real World Registry
Acronym: PIONEER
Status: Recruiting | Type: Observational
Sponsor: Mirai Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-21-001
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Skin Cancer; Gastrointestinal Cancer
Keywords: Pulsed Electric Fields; Reversible Electroporation; Electrochemotherapy; Ca-Electroporation
MeSH Terms: conditions — Skin Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry aims to assess real-world long-term disease outcomes for patients treated using reversible electroporation and a chemotherapeutic or calcium; in particular tumour response rates and recurrence rates. The study also aims to characterise side effects and the occurrence of Adverse Events and their relationship to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has been treated using Calcium Electroporation
* Any patient who has been treated using Electrochemotherapy
* Patients must be mentally capable of understanding the information given
* Patients must give written informed consent.

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study is a single arm, observational medical device registry designed to establish the efficacy and safety of treating solid tumours with reversible electroporation. ePORE, CUTIS and EndoVE are CE marked and are currently being used in the treatment of patients with solid tumours. This medical device registry will enable the collection of anonymised data which will enable the analysis and publication of high quality data to continuously support the efficacy and safety of these devices.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2036-06-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (CTCAE) | 5 years
  Safety evaluation will be performed via continuous assessment of safety parameters by reviewing events as they arise. The investigation will be put on hold if unacceptable safety issues are outstanding.
  Adverse Events (AE) and Serious Adverse Events (SAE) will be evaluated and graded according to Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Response Evaluation Criteria in Solid Tumours (RECIST) | 3 months, 12 months, 3 years, 5 years
  A response evaluation will be conducted at standard of care follow up

CONTACTS AND LOCATIONS:
Overall Officials: SEAN H Kinsella, Study Director — Mirai Medical
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT04929912/ICF_000.pdf